CLINICAL TRIAL: NCT00145249
Title: A Phase II Randomized Trial of Amphotericin B Alone or Combined With Fluconazole in the Treatment of AIDS-Associated Cryptococcal Meningitis
Brief Title: Amphotericin Alone or in Combination With Fluconazole for AIDS-Associated Meningitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-154; BAMSG 3-01
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Results first posted 2010-06-23 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2009-10

CONDITIONS: Cryptococcal Meningitis
Keywords: Bacterial infections, HIV infection, cryptococcal meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal; Bacterial Infections; HIV Infections | interventions — Amphotericin B; Fluconazole

ARMS (3):
- Standard Therapy (Active Comparator): Amphotericin B 0.7 mg/kg for 14 day followed by fluconazole 400 mg daily for 8 weeks. For subjects in the standard therapy arm whose Amphotericin B dose is continued beyond 14 days, fluconazole initiation will be delayed.
  Interventions: Drug: Amphotericin B; Drug: Fluconazole
- Fluconazole Low Dose (Experimental): Amphotericin B 0.7 mg/kg and the randomized dose of fluconazole at 400 mg/day for the first 14 days, then the randomized dose of fluconazole at 400 mg/day respectively for an additional 8 weeks.
  Interventions: Drug: Amphotericin B; Drug: Fluconazole
- Fluconazole High Dose (Experimental): Amphotericin B 0.7 mg/kg and the randomized dose of fluconazole at 800 mg/day for the first 14 days, then the randomized dose of fluconazole at 800 mg/day respectively for an additional 8 weeks.
  Interventions: Drug: Amphotericin B; Drug: Fluconazole

INTERVENTIONS:
Drug: Amphotericin B — Amphotericin B 0.7 mg/kg IV for the first 14 days of treatment. This period may be extended up to an additional 7 days.
Drug: Fluconazole — Fluconazole 400 or 800 mg daily. Among subjects whose baseline weight is less than 40 kg, randomized fluconazole doses will be 200 mg/kg daily or 400 mg/kg daily.

SUMMARY:
This study will examine the effectiveness and safety of a combination treatment for cryptococcal meningitis, a fungal infection common in persons with acquired immune deficiency syndrome (AIDS) in the developing world. The standard initial treatment includes two medications: amphotericin B for 2 weeks followed by 8 weeks of fluconazole. This study will look at whether study participants recover more quickly and have fewer side effects if they are given both drugs at the same time for 2 weeks followed by 8 weeks of fluconazole as compared to the standard treatment. Participants will be followed for approximately 6 months from the time they are enrolled into the study.

DETAILED DESCRIPTION:
This study is designed to address the need for more effective antifungal therapy for cryptococcal meningitis. This is a prospective, randomized, open-label, multicenter phase II clinical trial of combination therapy for the treatment of acute cryptococcal meningitis in HIV-positive subjects. The primary study objectives will be to assess the safety and tolerability of the study drug regimens; and to determine whether the safety and efficacy of combination therapy supports development of a phase III trial of combination therapy, and if so, to select the most appropriate dose of fluconazole plus amphotericin B based on safety and efficacy to be evaluated in a subsequent phase III trial. Secondary study objectives include: comparing the efficacy of the study drug treatments at 2, 6, and 10 weeks (Days 14, 42, and 70); comparing the findings on detailed neurological examination between study arms at baseline and 2, 6, 10, and 24 weeks (6 months); assessing the proportion of subjects in each study arm that are alive at 6 months after initiation of study therapy; describing the effects of baseline clinical, neurological, and mycological characteristics on mycological failure at 2 and 10 weeks; measuring time to cerebrospinal fluid (CSF) culture negatively for each study arm; assessing the length of hospitalization in the treatment groups as a surrogate of cost efficacy; assessing the incidence of immune reconstitution inflammatory syndrome among all subjects receiving highly active antiretroviral therapy (HAART); and examining antifungal susceptibility of all cryptococcal isolates. Study participants will include 150 subjects ages 13 and older. Subjects will be randomly assigned to 1 of 3 treatment arms including 1 standard therapy and 2 investigational arms. The standard treatment arm will include amphotericin B 0.7 mg/kg (IV) for 14 days followed by 8 weeks (56 days) of fluconazole at 400 mg/day orally. The 2 investigational arms will include daily amphotericin B 0.7 mg/kg (IV) and the randomized dose of fluconazole 400 mg/day or 800 mg/day for the first 14 day, then the randomized dose of fluconazole at 400 mg/day or 800 mg/day respectively for an additional 8 weeks (56 days). At the completion of study therapy, all subjects will receive chronic suppressive therapy with oral fluconazole at a dose of at least 200 mg/day. The safety endpoints are considered to be the primary endpoints for this study. The safety assessment for each treatment arm will end at study day 100 for each subject. The key safety endpoint will be the incidence of adverse experiences of grade 3-5 (total and attributed to the treatment regimens). The primary safety endpoint will examine the incidence of grade 3-5 adverse experiences that are definitely or probably related to study drugs, while secondary analysis will include grade 3-5 adverse experiences that are, definitely probably or possibly related to study drugs. Another secondary safety endpoint will be the number of dose-limiting toxicities attributed to the treatment regimens. Key efficacy endpoint (treatment success) will be a composite of the following 3 mycologic and clinical measures after 14, 42, and 70 days of therapy: CSF culture conversion; neurologically stable or improved; and alive. Other secondary efficacy endpoints that will be evaluated descriptively are: CSF culture conversion at multiple time points; all-cause mortality; length of hospitalization; and incidence of immune reconstitution inflammatory syndrome.

ELIGIBILITY:
Inclusion Criteria:

* First episode of cryptococcal meningitis as evidenced by a positive cerebrospinal fluid (CSF) stain or cryptococcal antigen, CSF culture pending
* Documentation of proven diagnosis of HIV-1 infection by acceptable labs at any time in the past: this testing includes Enzyme-linked immunosorbent assay (ELISA) or approved rapid testing method with confirmation by Western blot, a second positive ELISA, a positive HIV antigen, or HIV RNA detection.

OR

-Presumptive diagnosis of HIV-1 by approved rapid testing method at screening. This testing must be confirmed by a second ELISA (or Western blot), a positive HIV antigen, or HIV RNA detection within 10 days of study entry.

OR

* Presumptive HIV+. If serologic testing is not available, a history of an AIDS-defining illness (Category C, CDC, 1993) or any of the following conditions: extrapulmonary Pneumocystis carinii disease; multi-dermatomal herpes zoster (>10 lesions in a non-contiguous site); American trypanosomiasis (Chagas disease) of the CNS; Penicillium marneffei disease; visceral leishmaniasis; non-Hodgkin's lymphoma of any cell-type; Hodgkin's lymphoma; bartonellosis; microsporidiosis (>1 month's duration); nocardiosis; invasive aspergillosis; or Rhodococcus equi disease. Confirmation of HIV infection by lab testing, i.e., ELISA or approved rapid testing method with confirmation by Western blot, a second positive ELISA, a positive HIV antigen, or HIV RNA detection must be performed within 10 days of study entry.
* Subjects who are 13 years of age or greater.
* Baseline electrocardiogram (ECG) with QTc interval less than or equal to 500 milliseconds as determined by use of Fredericia's Correction formula.
* Ability of subject or legally authorized representative to give informed consent. For subjects who are unable to provide informed consent, sites will follow their own individual Institutional Review Board (IRB) policy regarding the informed consent process.

Exclusion Criteria:

* Pregnancy. Urine or serum testing must be performed at study entry or within the 7 days prior to study entry.
* Women of childbearing potential unwilling to use a medically approved and highly effective form of birth control while on study drug and for 2 weeks after last dose. Acceptable forms of birth control include an intrauterine device (IUD), oral contraceptives, condoms, abstinence, injectable contraceptive, or any other highly effective means of birth control. (A highly effective method of birth control is defined as those which result in a low failure rate [i.e. less than 1 percent per year] when used consistently and correctly.) Emergency contraceptive treatment and coitus interruptus are not considered effective forms of contraception.
* Breastfeeding.
* A concurrent central nervous system (CNS) process that in the opinion of the investigator would interfere with assessment of response, such as lymphoma, toxoplasmosis, or tuberculosis.
* Other conditions that in the opinion of the investigator would jeopardize the safety of a subject participating in the study or would render the subject unable to comply with the study plan, such as homelessness or IV drug use.
* Estimated creatinine clearance of less than 50 mL/min. NOTE: Testing must be performed at study entry or within the 7 days prior to study entry.
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 5x the upper limit of normal or bilirubin greater than 2.5 x the upper limit of normal. Results from tests performed within the 7 days prior to study entry may be used.
* Known intolerance of or allergy to fluconazole or amphotericin B.
* Subjects unlikely to survive for 2 weeks.
* Coma.
* More than 3 days of any systemic antifungal therapy for this fungal infection, or the need for concurrent systemic antifungal therapy, including flucytosine or interferon-g. Subjects taking fluconazole at less than or equal to 200 mg/day for prophylaxis are not excluded.
* Inability to take oral medications.
* Subjects who have received the following drugs within 7 days of study enrollment: rifampin, rifamycin, rifabutin, phenytoin, carbamazepine, cyclosporin A, tacrolimus, sirolimus, or long-acting barbiturates.
* Subjects who are receiving nevirapine at baseline.
* Strong clinical suspicion of untreated active tuberculosis. (Patients on anti-TB therapy not including rifampin or rifamycin may be eligible.)
* Previous participation in this study or ongoing participation in another trial with an investigational drug.
* Prior case of cryptococcosis with diagnosed central nervous system involvement.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2005-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (15):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - Harbor-UCLA Medical Center, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Harper University Hospital, Detroit, Michigan
  - Texas Medical Center - Michael E. DeBakey Veterans Affairs, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
- Thailand (5):
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Mahidol University - Siriraj Hospital - Medicine, Bangkok
  - Chiang Mai University, Chiang Mai
  - Khon Kaen University, Khon Kaen
  - Bamrasnaradura Institution, Nonthaburi

REFERENCES:
- [Result] Pappas PG, Chetchotisakd P, Larsen RA, Manosuthi W, Morris MI, Anekthananon T, Sungkanuparph S, Supparatpinyo K, Nolen TL, Zimmer LO, Kendrick AS, Johnson P, Sobel JD, Filler SG. A phase II randomized trial of amphotericin B alone or combined with fluconazole in the treatment of HIV-associated cryptococcal meningitis. Clin Infect Dis. 2009 Jun 15;48(12):1775-83. doi: 10.1086/599112. PMID 19441980
- [Result] Zimmer LO, Nolen TL, Pramanpol S, Wallace D, Walker ME, Pappas P, Chetchotisakd P. International collaboration between US and Thailand on a clinical trial of treatment for HIV-associated cryptococcal meningitis. Contemp Clin Trials. 2010 Jan;31(1):34-43. doi: 10.1016/j.cct.2009.11.002. Epub 2009 Nov 6. PMID 19897055

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 10 sites in the US and 5 sites in Thailand.
Groups:
- AmphoB Standard: Amphotericin B 0.7 mg/kg for 14 day followed by fluconazole 400 mg daily for 8 weeks. For subjects in the standard therapy arm whose Amphotericin B dose is continued beyond 14 days, fluconazole initiation will be delayed.
- AmphoB+Fluc400: Amphotericin B 0.7 mg/kg and the randomized dose of fluconazole at 400 mg/day for the first 14 days, then the randomized dose of fluconazole at 400 mg/day respectively for an additional 8 weeks.
- AmphoB + Fluc800: Amphotericin B 0.7 mg/kg and the randomized dose of fluconazole at 800 mg/day for the first 14 days, then the randomized dose of fluconazole at 800 mg/day respectively for an additional 8 weeks.
Period: Overall Study
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Started | 47 (47 subjects randomized; 45 subjects treated) | 48 (48 subjects randomized; 47 subjects treated-2 subjects randomized to AmphoB rec'd AmphoB+Fluc400) | 48 (48 subjects randomized; 49 treated-3 subjects randomized to AmphoB+Fluc400 rec'd AmphoB+Fluc800)
Completed | 36 | 33 | 31
Not Completed | 11 | 15 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800 | Total
Number analyzed (Participants) | 45 | 47 | 49 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 45 | 47 | 47 | 139
  >=65 years | 0 | 0 | 1 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 37.1 (8.47) | 36.5 (8.21) | 35.9 (9.44) | 36.5 (8.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 18 | 49
  Male | 29 | 32 | 31 | 92
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 14 | 42
  Thailand | 31 | 33 | 35 | 99

OUTCOME MEASURES:

1. Primary Outcome: Number of Grade 3-5 Adverse Experiences That Are Definitely or Probably Related to Study Drug
Description: Events are reported by MedDRA Preferred Term.
  Grade 3 - Severe. Incapacitating; inability to perform usual activities and daily tasks; significantly affects clinical status; requires therapeutic intervention.
  Grade 4 - Life-threatening. AE is life-threatening.
  Grade 5 - Death. AE causes death.
Time Frame: Day 100
Population: The Regulatory Safety population includes all subjects who were randomized, who receive at least 1 dose of study drug, and who have any on-study data.
Measure: Number; unit: Events
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 45 | 47 | 49
Events
  Hypomagnesaemia | 2 | 1 | 0
  Hypokalaemia | 0 | 0 | 1
  Anaemia | 1 | 1 | 0
  Drug intolerance | 1 | 0 | 0
  Creatinine renal clearance increased | 0 | 0 | 1
  Psychotic disorder | 0 | 0 | 1

2. Primary Outcome: Number of Dose-limiting Toxicities Attributed to Treatment Regimens
Description: Events are reported by MedDRA Preferred Term.
  Dose limiting toxicities include events that resulted in study drug being adjusted, interrupted, or discontinued.
Time Frame: Day 100
Population: as for outcome 1
Measure: Number; unit: Events
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 45 | 47 | 49
Events
  All Events | 6 | 7 | 14
  Blood creatinine increased | 4 | 1 | 1
  Creatinine renal clearance decreased | 0 | 1 | 2
  Creatinine renal clearance increased | 0 | 0 | 2
  Renal failure | 0 | 2 | 0
  Renal failure acute | 0 | 1 | 1
  Azotaemia | 0 | 0 | 1
  Renal impairment | 0 | 0 | 1
  Nausea | 0 | 0 | 1
  Vomiting | 0 | 0 | 1
  Drug intolerance | 1 | 1 | 0
  Chills | 0 | 1 | 0
  Neutropenia | 0 | 0 | 1
  Hepatitis acute | 1 | 0 | 0
  Pneumonia | 0 | 0 | 1
  Dehydration | 0 | 0 | 1
  Respiratory failure | 0 | 0 | 1

3. Secondary Outcome: Number of Deaths
Description: Number of deaths occurring on study.
  Day = Day relative to the first dose of study drug.
Time Frame: 14, 42, and 70 days
Population: The Regulatory Safety Population was used in this analysis, which includes all subjects who were randomized, who received at least 1 dose of study drug, and who have any on-study data.
Measure: Number; unit: Subjects
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 45 | 47 | 49
Subjects
  All Deaths | 10 | 8 | 9
  Day 1-14 | 3 | 2 | 1
  Day 15-42 | 3 | 2 | 1
  Day 43-70 | 1 | 2 | 5
  Day >70 | 3 | 2 | 2

4. Secondary Outcome: Number of Subjects With Cerebrospinal Fluid (CSF) Culture Conversion at Multiple Time Points
Description: Number of subjects that have a negative fungal culture at Baseline, Day 14, Day 42, and Day 70.
Time Frame: Baseline, 14, 42, and 70 days
Population: The modified Intent to Treat (mITT) population includes all subjects who are randomized to a treatment arm and receive any dose of study drug, who provide any outcome data, and who are determined to have met 2 key criteria for inclusion in the primary analysis - diagnosis of culture-proven cryptococcal meningitis and proven HIV infection.
Measure: Number; unit: Subjects
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 46 | 48 | 41
Subjects
  Baseline - Negative | 0 | 0 | 0
  Day 14 - Negative | 20 | 13 | 22
  Day 42 - Negative | 35 | 37 | 36
  Day 70 - Negative | 36 | 39 | 38

5. Secondary Outcome: Number of Subjects Meeting the Key Efficacy Endpoint of Treatment Success
Description: Treatment success is defined as a composite of the 3 mycologic and clinical measures: CSF culture conversion; neurologically stable or improved; and alive
Time Frame: 14, 42, and 70 days
Population: The mITT population includes all subjects who are randomized to a treatment arm and receive any dose of study drug, who provide any outcome data, and who are determined to have met 2 key criteria for inclusion in the primary analysis - diagnosis of culture-proven cryptococcal meningitis and proven HIV infection.
Measure: Number; unit: Subjects
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 46 | 48 | 41
Subjects
  Day 14 - Success | 19 | 13 | 22
  Day 42 - Success | 33 | 35 | 33
  Day 70 - Success | 33 | 36 | 32

6. Secondary Outcome: Number of Subjects Reporting Immune Reconstitution Inflammatory Syndrome (IRIS)
Description: Number of subjects reporting immune reconstitution inflammatory syndrome (IRIS) following treatment.
  Day = Day relative to first dose of study drug
Time Frame: 14, 42, and 70 days
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 45 | 47 | 49
Subjects
  Day 1 through 70 | 2 | 0 | 1
  Day 1-14 | 0 | 0 | 0
  Day 15-42 | 1 | 0 | 0
  Day 43-70 | 1 | 0 | 1

7. Secondary Outcome: Mean Days of Hospitalization
Description: Mean days of hospitalization. Includes days subject was hospitalized prior to study enrollment for current hospital stay.
Time Frame: 7, 14, 42, and 70 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 46 | 48 | 41
Days
  Day 7 | 8.9 (1.61) | 8.8 (2.39) | 8.1 (2.53)
  Day 14 | 15.4 (1.78) | 15.1 (3.27) | 13.6 (4.37)
  Day 42 | 16.3 (4.22) | 17.4 (5.91) | 16.5 (7.03)
  Day 70 | 16.7 (4.54) | 20.1 (11.63) | 16.6 (8.24)

8. Secondary Outcome: Number of Cryptococcal Isolates With Antifungal Susceptibility
Description: Isolates were collected at days 14 and 70 for assessment of antifungal susceptibility.
Time Frame: Days 14 and 70
Population: The study team has since determined that the assay that was to be utilized did not have sufficient sensitivity/specificity for its intended purpose and therefore these results will not be generated.
Measure: Number; unit: Isolates
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Mean Change in Neurological Exam Score From Baseline - Day 14
Description: Neurological assessment by Mini-mental Status Exam (MMSE). This is collected as a continuous variable with values from 0-30; where lower scores indicate greater impairment.
Time Frame: Baseline and Day 14
Population: The number of subjects tested in the modified Intent to Treat (mITT) population includes all subjects who are randomized to a treatment arm & receive any dose of study drug, who provide any outcome data, & who are determined to have met 2 key criteria for inclusion in the primary analysis: diagnosis of cryptococcal meningitis & HIV infection.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 40 | 43 | 40
Scores on a scale | 0.5 (4.07) | 2.1 (3.74) | 3.5 (6.25)

10. Secondary Outcome: Mean Change in Neurological Exam Score From Baseline - Day 42
Description: as for outcome 9
Time Frame: Baseline and Day 42
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 37 | 39 | 37
Scores on a scale | 1.6 (2.58) | 1.8 (4.42) | 3.3 (7.9)

11. Secondary Outcome: Mean Change in Neurological Exam Score From Baseline - Day 70
Description: as for outcome 9
Time Frame: Baseline and Day 70
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 37 | 34 | 30
Scores on a scale | 1.5 (3.28) | 2.2 (3.58) | 4.2 (6.84)

12. Secondary Outcome: Mean Change in Neurological Exam Score From Baseline - Day 168
Description: as for outcome 9
Time Frame: Baseline and Day 168
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Number analyzed (Participants) | 33 | 27 | 28
Scores on a scale | 2.0 (2.28) | 2.8 (3.92) | 4.4 (7.58)

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting on or after Day 0 and on or before Day 100.
Description: If a subject experienced more than 1 of a given AE, the subjects is counted only once for that AE. If a subject experienced more than one AE in a system organ class (SOC), the subject is counted only once in that SOC.
Arm/Group | AmphoB Standard | AmphoB+Fluc400 | AmphoB + Fluc800
Serious Adverse Events (participants affected / at risk) | 22/45 | 17/47 | 26/49
Other Adverse Events (participants affected / at risk) | 44/45 | 47/47 | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AmphoB Standard (N=45) | AmphoB+Fluc400 (N=47) | AmphoB + Fluc800 (N=49)
Sepsis (Infections and infestations) | 4 | 3 | 0
Meningitis cryptococcal (Infections and infestations) | 2 | 1 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 2
AIDS related complication (Infections and infestations) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
End stage AIDS (Infections and infestations) | 0 | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Toxoplasmosis (Infections and infestations) | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 3 | 2 | 2
Convulsion (Nervous system disorders) | 2 | 3 | 0
Headache (Nervous system disorders) | 1 | 1 | 1
Brain compression (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Hemiplegia (Nervous system disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Immune reconstitution syndrome (Immune system disorders) | 2 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
CSF pressure increased (Investigations) | 0 | 0 | 1
Prothrombin time prolonged (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papilloedema (Eye disorders) | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AmphoB Standard (N=45) | AmphoB+Fluc400 (N=47) | AmphoB + Fluc800 (N=49)
Hypokalaemia (Metabolism and nutrition disorders) | 38 | 38 | 39
Hypomagnesaemia (Metabolism and nutrition disorders) | 27 | 33 | 31
Anorexia (Metabolism and nutrition disorders) | 12 | 8 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 7 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 5 | 2 | 3
Vomiting (Gastrointestinal disorders) | 14 | 14 | 16
Nausea (Gastrointestinal disorders) | 4 | 14 | 16
Constipation (Gastrointestinal disorders) | 6 | 4 | 9
Diarrhoea (Gastrointestinal disorders) | 3 | 6 | 6
Anaemia (Blood and lymphatic system disorders) | 21 | 27 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 4 | 4
Sepsis (Infections and infestations) | 5 | 7 | 6
Herpes simplex (Infections and infestations) | 4 | 4 | 5
Sinusitis (Infections and infestations) | 7 | 0 | 6
Bacteraemia (Infections and infestations) | 1 | 3 | 5
Herpes zoster (Infections and infestations) | 3 | 4 | 1
Oral candidiasis (Infections and infestations) | 2 | 2 | 4
Pneumocystis jiroveci pneumonia (Infections and infestations) | 3 | 3 | 1
Headache (Nervous system disorders) | 10 | 13 | 14
Convulsion (Nervous system disorders) | 5 | 5 | 2
Intracranial pressure increased (Nervous system disorders) | 3 | 2 | 2
Phlebitis (Vascular disorders) | 4 | 5 | 8
Thrombophlebitis (Vascular disorders) | 2 | 4 | 6
Hypotension (Vascular disorders) | 4 | 2 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 4 | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 5
Insomnia (Psychiatric disorders) | 11 | 7 | 11
Pyrexia (General disorders) | 2 | 4 | 6
Chills (General disorders) | 4 | 4 | 2
Blood creatinine increased (Investigations) | 4 | 4 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 4 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 4 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 4
Hypertension (Vascular disorders) | 1 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 3
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Depression (Psychiatric disorders) | 0 | 0 | 3
Asthenia (General disorders) | 1 | 2 | 3
Pain (General disorders) | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Renal failure (Renal and urinary disorders) | 0 | 6 | 0
Papilloedema (Eye disorders) | 2 | 1 | 3
Immune reconstitution syndrome (Immune system disorders) | 3 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less